CLINICAL TRIAL: NCT01016366
Title: Randomised, Double Blind, Placebo Controlled Study of Lu AA24493 in Patients With Friedreich's Ataxia to Evaluate Safety and Tolerability and to Explore Efficacy
Brief Title: Safety Study of Carbamylated Erythropoietin to Treat Patients With the Neurodegenerative Disorder Friedreich's Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12631A; 2008-003662-25 (EudraCT Number)
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Friedreich's Ataxia
Keywords: Friedreich's Ataxia; FRDA; Neurodegenerative; Erythropoietin; Carbamylated; Neuroprotection; Frataxin
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lu AA24493 (Experimental)
  Interventions: Drug: Lu AA24493
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AA24493 — Vials with solution for i.v. injection. 325mcg Lu AA24493 dosed 3 times per week for two weeks. Vials will be supplied in concentrations ready for injection.
  Other Names: CEPO
  Arms: Lu AA24493
Drug: Placebo — Vials with solution for i.v. injection. Placebo dosed 3 times per week for two weeks.
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to determine whether carbamylated erythropoietin is a safe treatment for patients who suffer from Friedreich's Ataxia.

DETAILED DESCRIPTION:
Friedreich's Ataxia (FRDA) is a hereditary, progressive neurodegenerative disorder caused by mutations in the gene encoding frataxin. The mutation results in a severe reduction in levels of the mitochondrial protein, frataxin. A decline in frataxin levels and its associated consequences is believed to be the primary cause of symptoms in FRDA patients. The clinical symptoms of FRDA include progressive gait and limb ataxia, dysarthria, diabetes mellitus and hypertrophic cardiomyopathy. First symptoms usually appear between the age of 5 and 15 years. As the disease progresses the patient becomes confined to a wheel chair and at later stages the patients become increasingly incapacitated. There is currently no effective treatment for FRDA.

The naturally occurring hormone, erythropoietin (EPO), is able to protect various neuronal tissues from ischemic injury. Recombinant human erythropoietin (EPO) increases frataxin expression in lymphocytes from patients with FRDA. Also, EPO treatment of FRDA patients resulted in a favourable outcome compared to baseline as assessed by the levels of frataxin and biomarkers of oxidative stress. In a pilot study with EPO in FRDA patients, the treatment was well tolerated apart from the expected haematological (haematopoietic) side effects. Lu AA24493 (CEPO) is a modified (carbamylated) version of EPO, which is neuroprotective but without the haematopoietic side effects. Lu AA24493 is being developed for treatment of patients with FRDA.

Although the target for the non-haematological effects of Lu AA24493 (and EPO) is currently unknown, Lu AA24493 (CEPO) can protect cells and tissue from various types of injuries. Furthermore, in vitro Lu AA24493 (CEPO) increases the frataxin levels in lymphocytes from FRDA patients as well as from control patients. This study aims to evaluate the safety of 2 weeks treatment (6 doses, 3 doses per week) of CEPO in patients with FRDA and to explore efficacy by using neurological rating scales and by exploring levels of frataxin and biomarkers of oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been diagnosed with FRDA and has had a genetic test demonstrating >400 GAA nucleotide triplet repeats on the shorter of the two frataxin alleles
* The patient has a SARA (Stance) sub-score of <=6
* The patient has a SARA (Gait) sub-score of <=6
* Man or woman, aged 18 years or over
* If female then woman should agree not to try to become pregnant during the study, and use adequate protection/abstinence or not be of child bearing potential

Exclusion Criteria:

* Clinically significant unstable illnesses such as liver, kidney, heart, stomach problems unrelated to their disease of FRDA
* Disallowed medications
* Serious underlying disease
* Clinically significant abnormal vital signs unrelated to the underlying disease of FRDA
* Abnormal laboratory blood results considered by the doctor as clinically significant, e.g.anaemia
* Treatment with idebenone within 6 weeks prior to screening
* Treatment with erythropoietin within 16 weeks prior to screening
* Clinically significant abnormal ECG
* Received or donated blood within previous 3 months
* Participation within another clinical trial within past 30 days
* Pregnancy or breast feeding
* History of drug allergies or hypersensitivities
* Current (or within past 6 months) disorder related to drug or alcohol abuse (as defined DSM-IV-TR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of 2 weeks treatment with Lu AA24493 in patients with Friedreich's Ataxia | 2 week treatment phase + 4 week follow up period

SECONDARY OUTCOMES:
To explore biomarkers of efficacy, including frataxin, 8-OHdG & peroxides | 2 week treatment phase + 4 week follow up period
To explore efficacy by neurological assessment (Scale for the Assessment and Rating of Ataxia (SARA), Friedreich's Ataxia Rating Scale (FARS)) | 2 week treatment phase + 4 week follow up period
To explore efficacy by the Clinical Global Impression scales (CGI-I/S) | 2 week treatment phase + 4 week follow up period
To explore population pharmacokinetic parameters of Lu AA24493 | 2 week treatment phase + 4 week follow up period
To evaluate the immunogenicity of Lu AA24493 | 2 week treatment phase + 4 week follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (7):
- AT001, Innsbruck, Austria
- Germany (4):
  - DE004, Bochum
  - DE002, Bonn
  - DE001, Munich
  - DE003, Tübingen
- Italy (2):
  - IT001, Milan
  - IT002, Naples

REFERENCES:
- Available data/document: EMA EudraCT Results: 2008-003662-25 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2008-003662-25/results